CLINICAL TRIAL: NCT02408835
Title: A Randomised Controlled Trial Comparing PICO™ Single Use Negative Pressure Wound Therapy System (Smith & Nephew Healthcare Limited, UK) to Conventional Wound Care Following Inguinal Lymphadenectomy for Metastatic Cutaneous Malignancy
Brief Title: Negative Pressure Wound Therapy in Groin Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South Eastern Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Sandra McAllister, Academic Clinical Lecturer, South Eastern Health and Social Care Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPWT/14/1.0
Record Dates: First submitted 2014-12-19; First posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Neoplasm Metastasis; Secondary Malignant Neoplasm of Lymph Node; Non-healing Surgical Wound (Disorder); Skin Neoplasms
Keywords: negative pressure wound therapy; lymphadenectomy; wound healing
MeSH Terms: conditions — Neoplasm Metastasis; Lymphatic Metastasis; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICO™ (Active Comparator): Use of PICO™ system negative pressure wound therapy device on surgical wound for up to seven days.
  Interventions: Device: PICO™
- Conventional wound care (No Intervention): Usual wound dressings will be used as comparison group.

INTERVENTIONS:
Device: PICO™ — Negative pressure wound therapy device for closed surgical wounds.
  Other Names: PICO™, Smith & Nephew Healthcare, UK
  Arms: PICO™

SUMMARY:
This study investigates the use of a negative pressure wound therapy device (PICO™, Smith & Nephew Healthcare, UK) on clean, closed surgical wounds, in patients who are undergoing inguinal lymphadenectomy for metastatic carcinoma of cutaneous origin.

DETAILED DESCRIPTION:
Patients may develop inguinal lymph node metastases from a variety of cutaneous neoplasms. A number of factors conspire to cause a high rate of wound breakdown and other complications in this patient group. Reported rates of wound healing complications vary in the literature, but tend to affect > 40% of patients.

A new negative pressure wound therapy device is recommended for use in clean, closed surgical wounds (PICO™ system, Smith & Nephew Healthcare, UK). Patients will be randomised to receive either PICO™ system for up to seven days, or conventional dressings, and then assessed for wound healing and other outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-proven inguinal lymph node metastases from neoplasm of cutaneous origin

Exclusion Criteria:

* inability to give informed consent for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Time to wound healing | From date of surgery until epithelial integrity is restored at the surgical site. Assessed at least weekly until wound is healed, up to 20 weeks after surgery
  Determination of wound healing

SECONDARY OUTCOMES:
Wound infection As defined by Comprehensive Complication Index (CCI) | From date of surgery until wound is healed (epithelial integrity restored at surgical site), up to 20 weeks after surgery.
  As defined by Comprehensive Complication Index (CCI)
Lymphoedema (Limb volume measurements) | From date of surgery up to one year post-operatively.
  Limb volume measurements at 3, 6, 9 and 12 months
Need for further surgical interventions to achieve wound healing | From date of surgery until wound is healed, up to 20 weeks after surgery.
Scar appearance (POSAS) | From date of surgery up to one year post-operatively.
  POSAS at 3,6, 9 and 12 months
Patient reported outcomes (qualitative interview) | From date of surgery to six months post-operatively.
  Semi-structured qualitative interviews in first week after surgery, and at 6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hill, MB, Study Chair — South Eastern Health & Social Care Trust
Locations (1):
- The Ulster Hospital, Belfast, Northern Ireland, United Kingdom